CLINICAL TRIAL: NCT01374386
Title: RCMI Clinical Research Infrastructure Initiative: Exergaming
Brief Title: Impact of Exergaming on Adolescent Youth
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not receive funding.
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, David Martins, Professor of Medicine, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-10-2240-02
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Childhood Obesity
Keywords: adolescent obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Physical Activity (No Intervention): Participants in this arm are do not have access to Exergames, only usual physical activity at the gym
- Exergaming (Experimental): Participants in this arm will have access to usual physical activity at the gym as well as access to Exergaming equipment (video games that require physical activity)
  Interventions: Behavioral: Exergaming

INTERVENTIONS:
Behavioral: Exergaming — Participants will have access to Exergaming equipment (video games that require physical activity)
  Arms: Exergaming

SUMMARY:
The purpose of this study is to gather information on how much exercising with video games (ExerGaming) can increase the physical activity among overweight and youth. This study will try to see if participating in physical activity and exercising with video games at the same time can make overweight children move around more to better their own health. The hypothesis is that those in Exergaming arm will physiological changes and increase physical activity.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* aged 12-14 years
* baseline BMI > 25
* gender- and age-specific 85th percentile cutoff points from the CDC growth chart
* parental consent and subject assent

Exclusion Criteria:

* subjects not meeting the inclusion criteria or with physician-determined musculoskeletal, cardiopulmonary, metabolic, psychological, neuro-developmental or behavioral conditions that make mild-to-moderate physical activity potentially hazardous.
* Participants under the age of 12 are excluded from the study because Weingart YMCA has an age policy. Children under the age of 12 are not allowed to be at the facility alone. Therefore, the minimum age for the study is 12 years old so supervision is not a problem.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Change in mean daily physical activity | 2 years
  Change in mean daily physical activity from baseline (7-day activity log expressed as Kcal/day from relative MET intensity

SECONDARY OUTCOMES:
Change in caloric expenditure, body composition, and BMI | 2 years
  (a) Total daily caloric expenditure, (b) change in body composition (total body estimates of fat mass, fat-free mass, and lean body mass), and (c) change in BMI z score from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David Martins, MD, Msc, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States